CLINICAL TRIAL: NCT03914638
Title: Beta-agonist Efficacy and Tolerability as Adjuvant Therapy in Myasthenia Gravis
Acronym: BETA-MG
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Jan Lykke Scheel Thomsen, MD, PhD Fellow, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BETA-MG-01
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Albuterol; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Active intervention arm. Treatment for 8 weeks per treatment period.
  Interventions: Drug: Salbutamol 4Mg Tablet
- Placebo (Placebo Comparator): Placebo arm. Treatment for 8 weeks per treatment period.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Salbutamol 4Mg Tablet — Salbutamol 4 mg, three times daily
  Arms: Active
Drug: Placebo oral capsule — Placebo, three times daily
  Arms: Placebo

SUMMARY:
This study examines the effect of adjuvant therapy with the oral beta-agonist Salbutamol in patients with generalized myasthenia gravis on stable standard of care having residual symptoms.

DETAILED DESCRIPTION:
Myasthenia Gravis (MG) causes various degrees of increased muscular fatigue and ocular, bulbar, respiratory and extremity symptoms.

Residual symptoms often remain despite treatment with acetylcholinesterase inhibitors and immunosuppressive agents. Escalation of immunosuppressive treatment may provide additional benefit but is associated with potentially severe side effects, and high economic costs.

Treatment with beta-agonists has been investigated in animal models of MG, and in small, randomized pilot studies of generalized MG. Adjuvant therapy with oral beta-agonists in MG may be safe and cheap and may improve symptoms.

The trial will examine the tolerability and efficacy of adjuvant therapy with the oral beta-agonist Salbutamol in patients with generalized myasthenia gravis on stable standard of care having residual symptoms.

Present study is an investigator-initiated, randomized, placebo-controlled, rater and subject-blinded crossover study.

Study consists of Screening Period (4 weeks), Treatment Period 1 (8 weeks), Washout Period (4 weeks), Treatment Period 2 (8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Generalized myasthenia gravis (MGFA IIa-IVb) at screening, verified by ≥ 1 of the following: 1) AchR-antibodies in medical history, 2) Abnormal decrement on repetitive nerve stimulation in medical history
* Disease duration of ≥ 1 year
* Stable dose of antimyasthenic medications at screening
* Residual symptoms with a MG-QOL15 score of ≥ 10
* Age ≥ 18 years
* Ability to understand the requirements of the trial and provide written, informed consent

Exclusion Criteria:

* Evidence of malignancy ≤ 3 years prior to screening, unless deemed completely cured
* Thymectomy ≤ 6 months prior to screening
* Impending MG crisis or respiratory insufficiency
* Worsening of MG symptoms due to other diseases or medications (e.g. infection, beta-blockers, aminoglycosides, etc.)
* Other factor(s) or medical condition(s) that may explain residual symptoms
* Pregnancy or breast-feeding
* Treatment with beta-agonists
* Uncontrolled diabetes
* Ischemic Heart Disease, Cardiac Arrhythmia or Heart Failure (including hypertrophic cardiomyopathy)
* Uncontrolled Hypertension (≥ 160/110)
* Known hypersensitivity to any of the study drug components
* Treatment with tricyclic antidepressants, monoamineoxidase inhibitors, digoxine, or methylxanthines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Myasthenia Gravis Quality of Life 15-items (MG-QOL15) | 8 weeks (Treatment Period 1), 8 weeks (Treatment Period 2)
  Validated patient reported outcome-questionnaire consisting of 15 items and their impact on quality of life. Results are reported as change from baseline to 8 weeks of treatment in both treatment periods (Visit 4 compared to Visit 2, and Visit 7 compared to Visit 5).
Treatment Tolerability | 8 weeks (Treatment Period 1), 8 weeks (Treatment Period 2)
  Tolerability assessed by rate of adverse events and drug discontinuation in both treatment periods.

SECONDARY OUTCOMES:
Myasthenia Gravis Activity of Daily Living (MG-ADL) | 8 weeks (Treatment Period 1), 8 weeks (Treatment Period 2)
  Validated patient-reported outcome scale consisting of 8 disease-related items and their impact on activity of daily living. Results are reported as change from baseline to 8 weeks of treatment in both treatment periods (Visit 4 compared to Visit 2, and Visit 7 compared to Visit 5).
Neuro QOL | 8 weeks (Treatment Period 1), 8 weeks (Treatment Period 2)
  Patient reported fatigue-questionnaire used to rate fatigue and impact on quality of life. Results are reported as change from baseline to 8 weeks of treatment in both treatment periods (Visit 4 compared to Visit 2, and Visit 7 compared to Visit 5).
Quantitative Myasthenia Gravis (QMG) | 8 weeks (Treatment Period 1), 8 weeks (Treatment Period 2)
  Validated rating scale consisting of 13 items measuring muscle function and endurance. Results are reported as change from baseline to 8 weeks of treatment in both treatment periods (Visit 4 compared to Visit 2, and Visit 7 compared to Visit 5).
Myasthenia Gravis Composite (MG-Composite) | 8 weeks (Treatment Period 1), 8 weeks (Treatment Period 2)
  Validated scale consisting of 10 items with different weighting assessing severity of symptoms in MG. Results are reported as change from baseline to 8 weeks of treatment in both treatment periods (Visit 4 compared to Visit 2, and Visit 7 compared to Visit 5).

CONTACTS AND LOCATIONS:
Overall Officials: Jan LS Thomsen, MD, Study Director — University of Aarhus
Locations (2):
- Denmark (2):
  - Department of Neurology, Aalborg University Hospital, Aalborg
  - Neurology, Aarhus University Hospital, Aarhus

IPD SHARING:
Plan to Share IPD: No